CLINICAL TRIAL: NCT01135979
Title: Assessment of the Sympathetic Nervous System Blockade of the Upper Limb After a Brachial Plexus Block in Patients With End Stage Renal Failure
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 07AN007
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arterio-venous fistulae creation

SUMMARY:
The purpose of this study is to investigate what effect a local anesthetic nerve block of the arm in patients with end stage renal failure has upon blood flow in the skin of the arm.

DETAILED DESCRIPTION:
Aim

To quantify the degree of sympathetic blockade in the upper limb in patients with end stage renal failure produced during a regional anaesthetic technique, using laser Doppler flowmetry.

Hypothesis

Regional anaesthesia of the upper limb results in blockade of motor and sensory nerves, providing surgical and post-operative analgesia. Sympathetic nerves are also blocked resulting in local vasodilatation. This may be of benefit in surgery where enhanced blood flow is beneficial such as arterio-venous fistula creation. The degree and duration of sympathetic blockade produced by regional blocks however, has never been quantified. This study aims to quantify sympathetic blockade by measuring the changes in skin blood flow and skin temperature after placement of a brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal failure
* Over 18 years of age
* Written consent obtained
* Due to undergo surgery for forearm fistula creation under a regional block

Exclusion Criteria:

* Smokers
* Damaged skin on the arm
* Circulatory disorders such as Raynaud's disease, systemic sclerosis, sickle cell trait or disease
* Current use of beta blockers
* undergoing haemodialysis for more than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage renal failure who are due to have a forearm fistula created
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom